CLINICAL TRIAL: NCT04705688
Title: Platelet-activation and Optimal Inhibition in Patients With Atrial Fibrillation Undergoing Left Atrial Appendage Occlusion; The POPULAR-LAAO Trial
Brief Title: Platelet-activation and Optimal Inhibition in Patients With Atrial Fibrillation Undergoing Left Atrial Appendage Occlusion
Acronym: POPULAR-LAAO
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: R&D Cardiologie (Other)
Responsible Party: Principal Investigator, L.V.A. Boersma, Clinical professor, R&D Cardiologie
Other Study IDs: RDC-2020.02
Record Dates: First submitted 2020-12-22; First posted 2021-01-12 (Actual); Last update posted 2021-03-12 (Actual); Status verified 2021-03

CONDITIONS: Atrial Fibrillation
Keywords: Left atrial appendage occlusion; Device-related thrombus; Platelet reactivity; Coagulation activation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Biospecimen Retention: Samples With DNA — Blood samples will be preserved for analysis of hemostatic markers and CYP2C19 genotyping.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Left Atrial Appendage Occlusion: Patients undergoing left atrial appendage occlusion.

SUMMARY:
The POPULAR-LAAO registry is an open-label observational prospective registry to investigate hemostatic processes following left atrial appendage occlusion.

DETAILED DESCRIPTION:
This is an open-label observational prospective registry. The aim is to develop a better understanding of coagulation, platelet reactivity and prothrombotic factors in the first months after left atrial appendage occlusion, as occurrence of device-related thrombus and optimal postprocedural management remain a challenge after LAAO.

The study population will consist of patients with non-valvular atrial fibrillation (AF) at risk for cardio-embolic stroke scheduled for left atrial appendage occlusion. In these patients, blood samples for coagulation and platelet reactivity testing will be taken, which will be gathered prior to the procedure and 1 day, 14 days, 3 months and 6 months after the procedure. Data will be analyzed longitudinally and between groups based on patient characteristics.

ELIGIBILITY:
Inclusion Criteria:

* The subject is aged 18 years or older
* The subject is accepted/scheduled for left atrial appendage occlusion
* The subject has a CHA₂DS₂-VASc Score ≥2 (male) or ≥3 (female)
* The subject or legal representative is able to understand and is willing to provide written informed consent to participate in the trial.

Exclusion Criteria:

* Unable or unwilling to return for required follow-up visits and examinations
* Mechanical heart valves or valvular disease requiring surgery or interventional procedure
* Ongoing major bleeding or complicated or recent (<72hours) major surgery
* Known large oesophageal varices or decompensated liver disease (unless a documented positive opinion of a gastro-enterologist)
* Severe thrombocytopenia (<50,000/ml)
* High likelihood of being unavailable for follow-up or psycho-social condition making study participation impractical.
* Woman with child bearing potential who do not use an efficient method of contraception.
* Positive serum or urine pregnancy test for woman with child bearing potential
* Pregnancy or within 48 hours post-partum
* unsuitable LAA anatomy for occlusion or thrombus in the LAA at the time of procedure
* contraindications or unfavourable conditions to perform cardiac catheterization or transesophageal echocardiography (TEE)
* atrial septal malformations, atrial septal defect or a high-risk patent foramen ovale that may cause thrombo-embolic events
* atrial septal defect repair or closure device or a patent foramen ovale repair or any other anatomical condition as this may preclude an LAAO procedure
* Mitral valve regurgitation grade 3 or more
* Aortic valve stenosis (AVA<1.0 cm2 or Pmax>50 mmHg) or regurgitation grade 3 or more
* Planned carotid endarterectomy (CEA) for significant carotid artery disease
* Life expectancy of less than 1 year

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will consist of patients with non-valvular AF at high risk for cardio-embolic stroke scheduled for left atrial appendage occlusion.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2021-02-24 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Change in coagulation activation | Pre-LAAO and post-LAAO (1 day, 2 weeks, 3 months, 6 months)
  Influence of LAAO on coagulation activation over time
Change in platelet reactivity | Pre-LAAO and post-LAAO (1 day, 2 weeks, 3 months, 6 months)
  Influence of LAAO on platelet reactivity over time
CYP2C19 genotype | Pre-LAAO
  Rate of clopidogrel non-responders among LAAO patients will be assessed by determining CYP2C19 genotype

SECONDARY OUTCOMES:
Separate and composite event rates of stroke (ischemic or hemorrhagic), transient ischemic attack (TIA), systemic embolism and cardiovascular death. | Post-LAAO (3 months, 6 months, 12 months)
Major and minor bleeding event rate (according to Bleeding Academic Research Consortium criteria) | Post-LAAO (3 months, 6 months, 12 months)
Device related thrombus event rate | Post-LAAO (3 months, 12 months)

CONTACTS AND LOCATIONS:
Overall Officials: Lucas VA Boersma, MD PhD, Principal Investigator — St. Antonius Hospital
Locations (1):
- St. Antonius Ziekenhuis, Nieuwegein, Utrecht, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided